CLINICAL TRIAL: NCT04889612
Title: Analysis of the Influence of the Position of the Trunk and the Affected Upper Limb on Motor Coordination and Grip Strength of the Dominant and Non-dominant Hand and Wrist in Post-stroke Patients Compared to Healthy Controls.
Brief Title: Motor Coordination and Grip Strength of the Dominant and Non-dominant Hand and Wrist in Post-stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Olczak (Other)
Responsible Party: Sponsor-Investigator, Anna Olczak, PhD; Senior Specjalit of the Rehabilitation Clinc, Military Institute od Medicine National Research Institute
Organization: Military Institute od Medicine National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7/KRN/2019
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Stroke
Keywords: dominant hand; non-dominant hand; coordination; grip strength; stabilization; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- motor coordination and grip strength in dominant/non-dominant hand (Experimental): Dominant and non-dominant hand motor coordination and grip strength were tested in the stable position of the trunk and the upper arm, in post-stroke patients (study group) and in healthy subjects (control group).
  Interventions: Procedure: hand motor coordination in a sitting positin; Procedure: hand motor coordination in a supine position

INTERVENTIONS:
Procedure: hand motor coordination in a sitting positin — The subject sat on the therapeutic table (without back support), feet resting on the floor. The upper limb was to be examined in adduction of the humeral joint, with the elbow bent in the intermediate position between pronation and supination of the forearm, with free wrist and the hand. After putting the glove on, the subject was asked to make moves as quickly and in as full a range as possible. Finally, the measurement of grip strength with a dynamometer was performed.
Procedure: hand motor coordination in a supine position — In the supine position, the upper limb was stabilized at the subject's body (adduction in the humeral joint, elbow flexion in the intermediate position, wrist and hand free). After putting the Hand Tutor glove on, the subject was asked to make moves as quickly and in as full a range as possible. Finally, the measurement of grip strength with a dynamometer was performed.

SUMMARY:
This study aimed to assess how stabilization of the trunk and the upper extremity can change the parameters of hand/wrist motor coordination and grip strength in dominant and non-dominant paretic upper limb, in post-stroke patients and neurologically healthy subjects.

DETAILED DESCRIPTION:
The examination of the dominant and non-dominant paretic hand consisted of two motor tasks, carried out in two different starting positions: sitting and lying down (supine).

During the first examination, the subject sat on the therapeutic table (without back support), feet resting on the floor. The upper limb was examined in adduction of the humeral joint, with the elbow bent in the intermediate position between pronation and supination of the forearm, with free wrist and the hand.

In the supine position, the affected upper limb was stabilized at the subject's body (adduction in the humeral joint, elbow flexion in the intermediate position, wrist and hand free). The Hand Tutor device and an electronic hand dynamometer were used for the measurements. In each of the starting positions, after putting the glove on (using the Hand Tutor Device), the subject was asked to make moves as quickly and in as full a range as possible. Finally, the measurement of grip strength with a dynamometer was performed in both analyzed starting positions, after completing the range of motion and frequency tests.

ELIGIBILITY:
Stroke Inclusion Criteria:1) participants with ischemic stroke; 2) participants with hemiparesis after 5 to 7 week after stroke; 3) participants with stable trunk (the Trunk Control Test 70-100 points); 4) participants who were in a functional state allowing movements of the upper extremity (FMA-UE 40-66 motor function points); 5) muscle tension (MAS 0 -1+); 6) no severe deficits in communication, memory, or understanding what can impede proper measurement performance; Stroke Exclusion Criteria:1) stroke up to two weeks after the episode, 2) acute polyneuropathy and damage to peripheral nerves, 3) lack of trunk stability, 4) no wrist and hand movement, 5) muscle tension (˃2 MAS), 6) high or very low blood pressure, 7) dizziness, a malaise of the respondents.

Healthy Inclusion Criteria - 1) the control group consisted of participants free from the upper extremity motor coordination disorders; Healthy Exclusion Criteria: 1) participants with a history of neurologic or musculoskeletal disorders such as carpal tunnel syndrome, tendonitis, stroke, head injury, or other conditions that could affect their ability to active movement and grip hand; 2) with severe deficits in communication, memory, or understanding what can impede proper measurement performance;

Ages: 20 Years to 91 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Frequency of wrist movement (flexion to extension), cycles#/sec | up to 1 week
  The Hand Tutor allows measurements the speed or frequency (i.e., the number of cycles per second, where one cycle represents the movement from flexion to contraction).
Frequency of 1st, 2nd, 3rd, 4th, 5th finger movement (flexion to extension), cycles#/sec | up to 1 week
  The Hand Tutor allows measurements the speed or frequency (i.e., the number of cycles per second, where one cycle represents the movement from flexion to contraction).
Wrist maximum range of motion (ROM) [mm] | up to 1 week
  The Hand Tutor allows measurements of the maximum range of motion (ROM).
  ROM is a sum of the wrist flexion or extension angles (mm). ROM is a sum of all the finger flexion or extension angles (i.e. at the metacarpophalangeal (MCP), proximal interphalangeal (PIP), and distal interphalangeal (DIP) joints), mm.
1st, 2nd, 3rd, 4th, 5th finger maximum range of motion (ROM), [mm] | up to 1 week
  The Hand Tutor allows measurements of the maximum range of motion (ROM).
  ROM is a sum of the wrist flexion or extension angles (mm). ROM is a sum of all the finger flexion or extension angles (i.e. at the metacarpophalangeal (MCP), proximal interphalangeal (PIP), and distal interphalangeal (DIP) joints), mm.
Assessment of the grip strength | up to 1 week
  Grip strength, kg (a manual electronic dynamometer (EH 101) was used for grip strength measurement (error of measurement, 0.5 kg/lb)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Olczak, PhD, Principal Investigator — Rehabilitation Clinic, Military Institute of Medicine
Locations (1):
- Military Institute of Medicine, Warsaw, Masovian District, Poland

IPD SHARING:
Plan to Share IPD: No